CLINICAL TRIAL: NCT01363726
Title: Surveillance of Rotavirus Gastroenteritis Among Children <5 Years of Age Visiting the Pediatric Emergency Room in Southern Israel
Brief Title: Surveillance of Rotavirus Gastroenteritis in Children <5 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: pediatric infectious diseases unit,, Soroka U Medical center
Other Study IDs: sor415005ctil
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2005-10

CONDITIONS: Gastroenteritis; Rotavirus Infections
Keywords: surveillance Rotavirus Gastroenteritis Children; < 5 years of age; southern Israel; Signed informed concent
MeSH Terms: conditions — Gastroenteritis; Rotavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: Jewish and Bedouin children < 5 years of age in southern Israel

SUMMARY:
The purpose of this study is to monitor diarrheal disease and observe changes after the introduction of the rota vaccine.

DETAILED DESCRIPTION:
Monitoring of diarrheal disease and observe changes after the introduction of the rota vaccine Comparing the epidemiology in Jewish and Bedouin population before and after the introduction of the rota vaccine into the national immunization program

ELIGIBILITY:
Inclusion Criteria:

1. Children < 5 years with
2. Gastro enteritis
3. Visiting the ER
4. Residents of southern Israel
5. Signed informed concent -

Exclusion Criteria:

Not all of the above

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Survieillance of Rotavirus Gastroenteritis Among Children Bedouin and Jewish < 5 years with gastro enteritis visiting the ER in southern Israel
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2005-10

PRIMARY OUTCOMES:
epidemiology of rota virus disease in southern Israel before and after the rota virus vaccine introduction | 7 years
  To assess the proportion of rotavirus gastroenteritis among children <5 years of age visiting the pediatric ER in southern Israel. To assess the hospitalization rate due to rotavirus.

SECONDARY OUTCOMES:
To compare rotavirus gastroenteritis among children <5 years of age from Jewish and Bedouin populations. | 7 years
  To compare rotavirus gastroenteritis among children <5 years of age from Jewish and Bedouin populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric infectious disease unit Soroka U medical center, Beersheba, Israel